CLINICAL TRIAL: NCT00710905
Title: Visual Function With Contralateral AcrySof® ReSTOR® Aspheric SN6AD1 and SN6AD3
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Postmarket study terminated as the SN6AD3 is no longer promoted.
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCONsur002.08
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Cataract
Keywords: Cataract IOL ReSTOR Aspheric; Bilateral cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR (Experimental): Contralateral implantation of AcrySof ReSTOR +3 Intraocular Lens (IOL) in one eye, Acrysof ReSTOR +4 IOL in the other eye.
  Interventions: Device: AcrySof ReSTOR Aspheric IOL models SN6AD1 and SN6AD3

INTERVENTIONS:
Device: AcrySof ReSTOR Aspheric IOL models SN6AD1 and SN6AD3 — Contralateral implantation of AcrySof ReSTOR +3 Intraocular Lens (IOL) in one eye, AcrySof ReSTOR +4 IOL in the other eye following cataract removal.

SUMMARY:
The objective of this study is to prospectively evaluate the visual parameters in a series of patients after phacoemulsification cataract surgery in a series of patients bilaterally implanted with the AcrySof® ReSTOR® Aspheric Intraocular Lens (IOL) Models SN6AD1 And SN6AD3.

ELIGIBILITY:
Inclusion Criteria:

* Prospective subjects should be 21 years of age and older, be of any race and gender and meet study entry criteria. Subject must require extraction of cataracts followed by implantation of a posterior chamber intraocular lens (IOL). Subjects must be candidates for bilateral removal of the natural crystalline lens followed by implantation of a multifocal IOL and be willing and able to complete all follow-up visits.

Exclusion Criteria:

* Subjects with pre-existing conditions that could skew the results or are contraindications for the AcrySof® ReSTOR® IOL should be excluded from the study. Please consult the AcrySof® ReSTOR® Aspheric product inserts under "Precautions" for subject groups that should be excluded from this study.
* All subjects must have ≤ 0.75 diopters of astigmatism preoperatively as measured by Keratometry (K) readings. If the surgeon determines that a correction of cylinder is necessary postoperatively, this may be performed after the three month evaluations are completed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Blaylock, Principal Investigator
Locations (2):
- Canada (2):
  - Dr John Blaylock, Abbotsford, British Columbia
  - Dr Dominique Meyer, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject must require extraction of cataracts followed by implantation of a posterior chamber intraocular lens (IOL). Subjects must be candidates for bilateral removal of the natural crystalline lens followed by implantation of a multifocal IOL and be willing and able to complete all follow-up visits.
Period: Overall Study
Arm/Group | ReSTOR
Started | 50
Completed | 34
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 21
Gender [Number; unit: participants] — Gender information was not collected for one subject.
  participants
    Female | 24
    Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Binocular Visual Acuity at Near, Intermediate and Distance
Description: Binocular uncorrected and best corrected visual acuity (VA) was tested at 4 meters (m) (distance), 60 centimeters (cm) (intermediate), and near at preferred distance (distance chosen by each subject and recorded in cm; mean and standard deviation calculated) with a standard ETDRS chart for distance and a hand held chart for near. Scores were calculated using logMAR values. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better VA.
Time Frame: 6 months after surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | ReSTOR
Number analyzed (Participants) | 34
LogMAR
  Uncorrected distance VA (4 m) | 0.02 (0.08)
  Uncorrected intermediate VA (60 cm) | 0.31 (0.11)
  Uncorrected best near VA (34.11 cm +/- 4.23 cm) | -0.02 (0.10)
  Best corrected distance VA (4 m) | -0.04 (0.07)
  Best corrected intermediate VA (60 cm) | 0.31 (0.15)
  Best corrected best near VA (34.17 cm +/- 4.40 cm) | -0.01 (0.10)

ADVERSE EVENTS:
Time Frame: Surgical visit until 6 months after surgery.
Arm/Group | ReSTOR
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReSTOR (N=50)
Retinal Detachment (Eye disorders) | 1 (1) — non-fatal medical event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReSTOR (N=50)
Posterior Capsule Opacification (Eye disorders) | 4 (5)
Visual disturbances (Eye disorders) | 2 (2) — Visual disturbances including, but not limited to: floaters and flashes, photopsia
Allergic Reaction (Eye disorders) | 1 (1) — Mild allergic reaction to prednisolone eye drops
Redness (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
When a clinical study report or manuscript, in lieu of a final report, is completed, Alcon will provide the summary findings of the study to the investigator.